CLINICAL TRIAL: NCT04857801
Title: Teduglutide in Short Bowel Syndrome Patients - A Way Back to Normal Life?
Brief Title: Teduglutide in Short Bowel Syndrome Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Felix Harpain, Principle Investigator, Medical University of Vienna
Other Study IDs: 131290
Record Dates: First submitted 2021-04-19; First posted 2021-04-23 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — teduglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Teduglutide — effect of teduglutide on intestinal rehabilitation

SUMMARY:
A retrospective analysis was performed using data of patients suffering from non-malignant SBS-IF. They were treated with teduglutide in a multidisciplinary SBS-IF program at a single university medical center between June 2016 and June 2020.

ELIGIBILITY:
Inclusion Criteria:

* SBS-IF

Exclusion Criteria:

* < 18 years
* Incompliance
* < 6 months of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SBS-IF patients receiving teduglutide for at least 6 months
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
enteral autonomy | at least 6 months of teduglutide treatment
  percentage of patients reaching complete discontinuation of parenteral support

IPD SHARING:
Plan to Share IPD: No